CLINICAL TRIAL: NCT06983015
Title: The Effect of Sticky Bone vs Cross-linked Hyaluronic Acid With Xenograft in Socket Preservation: Randomized Controlled Trial
Brief Title: Sticky Bone vs Xenograft With Cross-linked Hyaluronic Acid in Socket Preservation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed Salah Ali Mohamed, oral and maxillofacial surgery master candidate, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: socket preservation
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Socket Preservation
Keywords: sticky bone; xenograft with cross-linked hyaluronic acid

STUDY DESIGN:
Intervention Model Description: This prospective randomized (1:1) blinded clinical trial used an unstratified random block design (block sizes2, 4, and 6) to ensure balance in the number of patients assigned to each group. Informed consent for sharing clinical data and images for scientific purposes will be collected from all patients prior to commencement of the study, which was performed in accordance with the Declaration of Helsinki.
  The patients will be randomly assigned to one of the two groups according to the graft material: group I (Sticky bone) and group II (cross linked hyaluronic acid mixed with xenograft) where each patient will received either sticky bone or cross linked hyaluronic acid mixed with xenograft in the extraction socket according to the treatment group by the same operator. The graft material for extraction socket will be the primary predictor variable.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sticky bone (Experimental): patients in this group will undergo tooth extraction and immediate augmentation using sticky bone
  Interventions: Procedure: sticky bone
- xenograft mixed with cross-linked hyaluronic acid (Active Comparator): patients in this group will undergo tooth extraction and immediate augmentation using xenograft mixed with cross-linked hyaluronic acid
  Interventions: Procedure: xenograft mixed with cross-linked hyaluronic acid

INTERVENTIONS:
Procedure: sticky bone — extraction socket will be augmented using a sticky bone.
  Arms: sticky bone
Procedure: xenograft mixed with cross-linked hyaluronic acid — Socket will be augmented with a mixture of xenograft and cross linked hyaluronic acid.
  Arms: xenograft mixed with cross-linked hyaluronic acid

SUMMARY:
The present study aimed to evaluate clinical and radiographic outcomes of sticky bone in comparison to crosslinked hyaluronic acid mixed with xenograft in alveolar ridge preservation.

DETAILED DESCRIPTION:
After teeth extraction, the alveolar process goes through a remodeling process that leads to dimensional changes that end up with a decrease in the width and height of the alveolar bone; these changes happening after tooth loss proves that the alveolar process bone is tooth dependent.

Alveolar bone remodeling is a physiological process observed after tooth extraction that may compromise the subsequent dental implant rehabilitation. Most of the alveolar bone loss occurs during the first 3-6 months after tooth extraction, resulting in a bone width loss of 29-63%, which leads to difficulties restoring the teeth either with conventional prosthesis or with implant supported prosthesis and in many cases implant placement becomes a challenge.

To compensate for this alveolar remodeling and create an aesthetically implantsupported prosthesis, many bone grafting techniques were proposed, including guided bone regeneration, onlay bone block, and alveolar ridge preservation.

The latter is a prophylactic technique that involves inserting various biomaterials into the socket to reduce post-extraction changes. The two most commonly used bone grafting materials are allografts and xenografts. The Alveolar ridge preservation seeks to achieve successful ridge reconstruction, which involves the production of new bone within the volume of the old socket. Although xenografts provide steady and adequate bone volume maintenance, their healing time and the percentage of de novo bone production remain their main downside.

To improve alveolar ridge preservation outcomes, researchers are attempting to reduce the healing period so that implants can be placed shortly after tooth extraction. As a result, numerous growth factors were investigated as biological adjuvants to aid in the healing process and prevent physiological post-extractive bone loss. Recent researches studied the use of cross-linked hyaluronic acid (xHyA) gel as a biological adjuvant to xenograft in order to increase regeneration capacity and decrease post-extraction resorption Hyaluronic acid an extracellular polymer of disaccharides administration appears to have a beneficial impact on the healing process and bone cell response by stimulating mesenchymal cells proliferation, growth factors attraction and angiogenesis in situ. the cross-linked hyaluronic acid had been introduced with a slow degradation profile to maintain a longer presence. The combination of crosslinked hyaluronic acid mixed with xenograft was proved to be better than the xenograft only regarding post-extraction socket bone regeneration "Sticky bone" is a composite biomaterial designed for bone regeneration, combining particulate bone substitutes with autologous platelet aggregates, such as PRF and concentrated growth factors. This adaptable material conforms to various bony defects, preventing graft movement and preserving bone volume during healing, thus minimizing the need for block bone and titanium mesh.

The sticky bone had been used in socket preservation and provides good bone quality for further implant placement. The placement of sticky bone resulted in grafted material adherence to the recipient sites without micro and macro movements, and the PRF matrix prevented early epithelial ingross onto the defect site, resulting in significant new bone gain in both horizontal and vertical dimensions Sareen et al. reported in their systematic review that a major limitation was the lack of randomized controlled trials that provide evidence on alveolar ridge preservation with sticky bone. They recommend larger studies to evaluate the interest of sticky bone in various surgical procedures by comparing it with other existing materials and conventional techniques.

The present study aimed to evaluate clinical and radiographic outcomes of sticky bone in comparison to crosslinked hyaluronic acid mixed with xenograft in alveolar ridge preservation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Patient with hopeless maxillary anteriors and premolar with cl ii socket that needs extraction and delayed implant placement.

Exclusion Criteria:

* Acute abscesses or active infections localized in the proximity of the surgical field.
* Presence of heavy metallic artefacts that can distort CBCT scans
* Bad oral hygiene and non-compliance.
* Systemic diseases interfering with bone healing.
* Active and progressive periodontal disease
* Smoking, alcoholism and drug abuse
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
A standardized region of interest (ROI) will be calibrated for all sites, determined by following reference points | This measurement will be obtained at immediate postoperative and 6-months postoperative.
  A standardized region of interest (ROI) will be calibrated for all sites, determined by following reference points (8):
  * Apico-coronally: Coronally the most crestal bone peak will be detected mesially and distally; apically, an artificial line was drawn 1.5 mm below the most apical point of the root tip across the apical base of the socket.
  * Mesio-distally: limited by an artificial line at 1.5 mm distance of the most mesial and distal surface of adjacent tooth or implant.
  * Bucco-lingually: limited to the mostly detectable bone width extension.

SECONDARY OUTCOMES:
Bone density | This measurement will be obtained at immediate postoperative and 6-months postoperative.
  Bone density: this will be measured immediately postoperative and at 6- monthpostoperative interval
Postoperative Pain | at the following intervals: 1, 3, 7th day postoperative.
  Postoperative Pain: will be assessed using pain score for assessment of quality of life measured on a 10-point visual analogue scale (VAS), the 0 indicating no pain and 10 indicating the worst pain ever at the following intervals: 1, 3, 7th day postoperative.
Bone volume | This measurement will be obtained at immediate postoperative and 6-months postoperative.
  Bone volume: alveolar ridge volumetric change, pre- and postoperative CBCT scans will be superimposed. In order to calculate the volumetric resorption rate (Percentage)